CLINICAL TRIAL: NCT06510075
Title: Providing an Optimized and emPowered Pregnancy for You (PᵌOPPY) Aim 3: Randomized Controlled Trial
Brief Title: Providing an Optimized and Empowered Pregnancy for You (POPPY) Aim 3: Randomized Controlled Trial
Acronym: P3OPPY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Heart Association (Other); ConnectionHealth (Unknown); Memora Health (Unknown)
Responsible Party: Principal Investigator, Rachel Sinkey, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 300013085; 22HERNPMI985239 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Complications; Maternal Distress; Adverse Birth Outcomes; Infant Conditions
Keywords: Pregnancy outcomes; Health inequities
MeSH Terms: conditions — Pregnancy Complications | interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: Study is a randomized trial (n=400) randomizing eligible participants to usual care (n=100), or usual care plus a digital health intervention (n=100), or usual care plus a community health worker intervention (n=100), or usual care plus both a digital health intervention and a community health worker intervention (n=100).
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Digital Health Intervention (DHI) (Experimental): This group will receive routine prenatal care services. Additionally, those randomized to this arm will receive a DHI intervention. A modified DHI will be utilized that was developed by Memora Health in conjunction with EQUATE partners at UPenn and feedback from the POPPY Study Team and Community Advisory Board. All content is designed for 7th grade Flesch-Kincaid level or lower.
  Interventions: Behavioral: Digital Health intervention
- Community health worker (CHW) (Experimental): Individuals randomized to this group will receive routine prenatal care services. Additionally, they will receive a CHW intervention. The CHW intervention will be adapted from an ongoing CHW program in Jefferson County, AL called "From Day One (FDO)", a comprehensive patient-centered program designed to educate and provide non-clinical, psychosocial, emotional support to expectant mothers from the 1st trimester of pregnancy through 12 weeks postpartum. The intervention has been modified by the POPPY Study Team and Community Advisory Board
  Interventions: Behavioral: Community Health Worker
- DHI Plus CHW (Experimental): This group will receive routine prenatal care services. Additionally, this group will receive both DHI and CHW interventions.
  Interventions: Behavioral: Digital Health Intervention plus Community Health Worker
- Usual Care (No Intervention): This group will receive routine prenatal care services.

INTERVENTIONS:
Behavioral: Digital Health intervention — Health care information delivered via a link in a text message that is then opened in a secure browser.
  Other Names: DHI
  Arms: Digital Health Intervention (DHI)
Behavioral: Community Health Worker — Health care information delivered via CHW.
  Other Names: CHW
  Arms: Community health worker (CHW)
Behavioral: Digital Health Intervention plus Community Health Worker — Health care information delivered via DHI plus CHW
  Other Names: DHI plus CHW
  Arms: DHI Plus CHW

SUMMARY:
The PᵌOPPY study is designed to support the American Heart Association's mission to improve maternal/infant health outcomes and address inequities in maternal/infant health care. The P3OPPY Project is one of five projects within the American Heart Association P3 EQUATE Network. The overarching goal of the P3 EQUATE American Heart Association Health Equity Research Network (HERN) is to promote equity in Maternal and Infant Health outcomes by identifying innovative and cost-effective strategies to enhance access to quality health information, care, and experiences during pregnancy, postnatal and postpartum/preconception periods, particularly for Black and under-served populations. Collectively, the investigators will collaborate with pregnant and postpartum individuals and their families, hospitals, and communities to discover ways to reduce racism and social problems that contribute to poor health outcomes. In this trial, 400 non-Hispanic Black participants will be randomized to see if 2 promising interventions (digital health interventions and community health workers) reduce adverse pregnancy outcomes.

DETAILED DESCRIPTION:
The aim of this trial is to assess whether an existing Digital Heath Intervention (DHI) and/or a Community Health Worker (CHW) Intervention will reduce adverse maternal and perinatal outcomes. A 2 x 2 factorial randomized controlled trial of Non-Hispanic Black (NHB) patients living in high area deprivation index (ADI) communities will be conducted. Participants (n=400) will be randomized 1:1:1:1 to one of 4 arms: 1) standard prenatal care (PNC) alone, or 2) standard PNC plus DHI, or 3) standard PNC plus CHW, or 4) standard PNC, plus DHI and CHW.

The PᵌOPPY study is designed to support the American Heart Association's mission to improve maternal/infant health outcomes and address inequities in maternal/infant health care. The promise of digital health and community health worker engagement makes PᵌOPPY interventions potentially transformative, sustainable, and scalable for Non-Hispanic Black mothers and their infants from under-served communities in Alabama and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Self Identifies as Non-Hispanic Black
* Between 16-49 years old
* Pregnant individuals between 8⁰ - 22⁶ weeks gestational age
* Live singleton or dichorionic twin gestation
* Dating sonogram at <23 weeks gestation,
* Area Deprivation Index (ADI) National 4th or 5th Quintile
* Planning to deliver at UAB Hospital
* Speaks and writes in English
* No indication for delivery at the time of enrollment

Exclusion Criteria:

* Declines randomization
* Speaks or writes in languages other than English
* Currently incarcerated
* Fetal demise diagnosed prior to enrollment
* Known major structural chromosomal abnormalities prior to enrollment
* Participated in POPPY Pilot

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Weighted Adverse Outcome Score (WAOS) | [Time Frame: From randomization to 6 weeks postpartum]
  WAOS, calculated by adding the weights of all adverse events divided by the total number of deliveries.
  Maternal death=750, Neonatal death=400, Uterine rupture=100, Maternal ICU Admission=65, Birth trauma=60, Unanticipated operative procedure=40, NICU Admission=35, 5-minute Apgar <7=25, Maternal blood transfusion=20, and 4th degree perineal lacerations=5.

SECONDARY OUTCOMES:
Outpatient Prenatal Care Visits | Duration of pregnancy through 6 weeks postpartum
  Number of outpatient prenatal care and postpartum visits
Preterm Birth | At birth
  Delivery of a neonate at less than 37 weeks
Neonatal birthweight | At birth
  Weight of neonate at birth
Cesarean delivery | At birth
  Occurrence of a cesarean birth
Maternal blood transfusion | Duration of pregnancy through 6 weeks postpartum
  Transfusion of blood products
Breastfeeding intent | From randomization to delivery of the infant(s)
  Participant's self-reported intent of whether or not to express breast milk upon admission to the delivery-associated hospitalization
Maternal postpartum readmission | From discharge from the delivery-associated hospitalization to 6 weeks postpartum
  Admission of the mother to the hospital after discharge from the delivery-associated hospitalization
Neonatal hospital readmission | Birth to 6 weeks of life
  Admission of a neonate to the hospital after discharge from the hospital after birth

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Sinkey, MD, Principal Investigator — University of Alabama at Birmingham; Wally Carlo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No